CLINICAL TRIAL: NCT04253158
Title: Drug and Alcohol Prevention for College Athletes
Brief Title: Implementation of a Web-based Alcohol and Other Drug Prevention Intervention for Collegiate Student-athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prevention Strategies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1011
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Alcohol Drinking; Social Norms; Expectations; Harm Reduction
MeSH Terms: conditions — Alcohol Drinking; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Educational standard (Experimental): The aim of this arm is to increase knowledge about alcohol and other drug use.
  Interventions: Behavioral: Educational standard
- Educational standard and Harm prevention (Experimental): The aim of this arm is to increase knowledge about alcohol and other drug use and increase intentions for the use of harm prevention strategies.
  Interventions: Behavioral: Educational standard and Harm prevention
- Educational standard and Expectancies (Experimental): The aim of this arm is to increase knowledge about alcohol and other drug use and shift alcohol-related expectancies.
  Interventions: Behavioral: Educational standard and Expectancies
- Expectancies and Harm prevention (Experimental): The aim of this arm is shift alcohol-related expectancies and increase intentions to use harm prevention strategies.
  Interventions: Behavioral: Expectancies and Harm prevention
- Educational standard and Normative perceptions (Experimental): The aim of this arm is to increase knowledge about alcohol and other drug use and correct erroneous alcohol-related normative perceptions.
  Interventions: Behavioral: Educational standard and Normative perceptions
- Normative perceptions and Harm prevention (Experimental): The aim of this arm is to correct erroneous alcohol-related normative perceptions and increase intentions to use harm prevention strategies.
  Interventions: Behavioral: Normative perceptions and Harm prevention
- Educational standard, Normative Perceptions, and Expectancies (Experimental): The aim of this arm is to increase knowledge about alcohol and other drug use, correct erroneous alcohol-related normative perceptions, and shift alcohol-related expectancies.
  Interventions: Behavioral: Educational standard, Normative Perceptions, and Expectancies
- Normative perceptions, Expectancies, and Harm Prevention (Experimental): The aim of this arm is to correct erroneous alcohol-related normative perceptions, shift alcohol-related expectancies, and increase intentions to use harm prevention strategies.
  Interventions: Behavioral: Normative perceptions, Expectancies, and Harm Prevention

INTERVENTIONS:
Behavioral: Educational standard — Behavioral intervention aimed at increasing knowledge about alcohol and other drugs.
  Arms: Educational standard
Behavioral: Educational standard and Harm prevention — Behavioral intervention aimed at increasing knowledge about alcohol and other drugs increasing intentions to use harm prevention strategies.
  Arms: Educational standard and Harm prevention
Behavioral: Educational standard and Expectancies — Behavioral intervention aimed at increasing knowledge about alcohol and other drugs and shifting alcohol-related expectancies.
  Arms: Educational standard and Expectancies
Behavioral: Expectancies and Harm prevention — Behavioral intervention aimed at correcting erroneous norms about alcohol use and shifting alcohol-related expectancies.
  Arms: Expectancies and Harm prevention
Behavioral: Educational standard and Normative perceptions — Behavioral intervention aimed at increasing knowledge about alcohol and other drugs and correcting erroneous norms about alcohol use.
  Arms: Educational standard and Normative perceptions
Behavioral: Normative perceptions and Harm prevention — Behavioral intervention aimed at correcting erroneous norms about alcohol use and increasing intentions to harm prevention strategies.
  Arms: Normative perceptions and Harm prevention
Behavioral: Educational standard, Normative Perceptions, and Expectancies — Behavioral intervention aimed at increasing knowledge about alcohol and other drugs, correcting erroneous norms about alcohol use, and shifting alcohol-related expectancies.
  Arms: Educational standard, Normative Perceptions, and Expectancies
Behavioral: Normative perceptions, Expectancies, and Harm Prevention — Behavioral intervention aimed at correcting erroneous norms about alcohol use, shifting alcohol-related expectancies, and increasing intentions to use harm prevention strategies.
  Arms: Normative perceptions, Expectancies, and Harm Prevention

SUMMARY:
The broad aim of the proposed study is to use the innovative Multiphase Optimization Strategy to develop a highly effective Internet-delivered intervention, myPlaybook, for the prevention of substance use among college student-athletes. myPlaybook will undergo two rounds of randomized experimentation and targeted revision. At the conclusion of the second round, the optimized version of myPlaybook will be evaluated in large-scale Randomized Controlled Trial (RCT).

DETAILED DESCRIPTION:
College student-athletes are at increased risk of heavy alcohol use, smokeless tobacco use, and the use of performance enhancing substances as compared to non-athlete college students. Despite recent research underscoring the need for athlete-tailored interventions, there are no evidence-based options for the prevention of substance use among college student-athletes that take into account their unique patterns and motivations for use. This void leaves colleges with few easy-to-use, effective, and economical options for meeting the needs of their student-athletes and the minimum drug education requirements set by their governing organizations. The broad aim of the proposed study is to use the innovative Multiphase Optimization Strategy to develop a highly effective Internet-delivered program (myPlaybook) for the prevention of substance use among college student-athletes. The MOST approach is a systematic method for making decisions about program development and adaptation that are based on the performance of individual program components. The five core lessons of myPlaybook will undergo two rounds of randomized experimentation and targeted revision. At the conclusion of the second round, the newly optimized version of myPlaybook will be assembled and evaluated in large-scale Randomized Controlled Trial (RCT). This "beta" version of myPlaybook will be compared to an Internet-based college alcohol intervention with proven effectiveness with general college students. This approach will allow us to 1) develop an intervention that is optimized for considerable impact on substance use outcomes and 2) demonstrate the need for interventions specifically adapted for college student-athletes. The proposed research will be among the first demonstrations of the MOST approach for building and evaluating behavioral interventions with greatly enhanced public health impact. PUBLIC HEALTH RELEVANCE: This project has the potential to contribute to the health and safety of the more than 460,000 college student-athletes in the US. A contribution to the science of prevention will be made by demonstrating an innovative approach for the development and revision of behavioral interventions that focuses on achieving both statistical significance and optimizing public health impact.

ELIGIBILITY:
Inclusion Criteria:

* equal to or greater than 18 years of age
* registered first year student-athlete
* competes on NCAA sponsored team
* full-time NCAA collegiate student-athlete

Exclusion

* equal to or less than 17 years of age
* greater than 25 years of age
* non-NCAA sponsored athlete

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3859 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Descriptive norms: DRINKING NORMS RATING FORM (adapted DNRF) | past 30-day
  This scale (0-100%) measured the perceptions about the frequency of others' alcohol use. Perceived weekly drinking was computed by summing the reported estimates of drinking for each day of the week for the typical student. The lower the score the better.
Injunctive norms:DRINKING NORMS RATING FORM (adapted DNRF) | past 30-day
  This scale (0-100%) measured the perceptions about the frequency of others' approval of alcohol use. Perceived approval of alcohol use of others was computed by summing the reported estimates of approval compared to the actual approval as reported by the typical student. A lower score on this scale results in more positive effects.
Negative expectancies: COMPREHENSIVE EFFECTS OF ALCOHOL Scale (adapted CEOA) | past 30-day
  This agreement scale (1-4) measured negative expectancies (e.g., consequences of risks and/or aggression) of alcohol related effects. Sub-scale scores are calculated as the sum of respective items. A lower score on this scale results in more positive effects.
Positive expectancies: COMPREHENSIVE EFFECTS OF ALCOHOL Scale (adapted CEOA) | past 30-day
  This agreement scale (1-4) measured positive expectancies (e.g., socialability) of alcohol related effects. Sub-scale scores are calculated as the sum of respective items. A higher score on this scale results in more positive effects.

SECONDARY OUTCOMES:
PROTECTIVE BEHAVIORAL STRATEGIES SCALE-20 (adapted - PBSS-20) | past 30-day
  Intentions to use protective behavioral strategies (e.g., alternating alcoholic and non-alcoholic drinks). This intentions scale (1-7) measured future intent to use alcohol-related harm prevention strategies (e.g., alternating alcoholic and non-alcoholic drinks). A higher score on this scale results in more positive effects.